CLINICAL TRIAL: NCT03570268
Title: Educational and Exercise Intervention to Prevent Falls and Participation Restrictions in Subjects With Neurological Diseases
Brief Title: Preventing Falls and Participation Restrictions in Neurological Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2010-2318552
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis; Parkinson Disease; Stroke
Keywords: Falls prevention; Education; Neurological disease
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease; Stroke; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Education group (Experimental): Participants in the experimental intervention group (education group) received an educational program and tailored home exercises. This intervention consist of multiple, interacting components supported by a handbook and audio-video material designed to teach people the skills, techniques, and strategies for preventing falls, and increase social participation and engagement in inactivity of daily living. . After the educational session, two one hour sessions were spent to teach safe balance exercises that were developed in preceding studies, the patient was invited to perform at home for 2 months.
  Interventions: Other: Experimental Group: Education
- Control Group: Usual care (Active Comparator): Participants allocated to the control group received ongoing usual treatments. In addition, two one hour lessons were spent to teach stretching exercises that the patient was invited to perform at home for 2 months.
  Interventions: Other: Control Group: Usual care

INTERVENTIONS:
Other: Experimental Group: Education — Participants in the experimental intervention group received an educational program and tailored home exercises.
  Arms: Experimental group: Education group
Other: Control Group: Usual care — Participants allocated to the control group received stretching exercises.
  Arms: Control Group: Usual care

SUMMARY:
A randomized open clinical trial to assess the added value of a comprehensive rehabilitation program on fall prevention and improve participation and activities of daily living. Baseline assessment, 6-month experimental intervention (experimental group) vs. usual rehabilitation programs and assessment at end of treatment and six months after treatment will be performed.

DETAILED DESCRIPTION:
90 patients will be randomly patients will be stratified by disease type and randomized separately.

The trial will be organized in Baseline assessment (clinical characteristics; fall predictors, chosen among the variables found to predict falls in the observational study), experimental intervention (experimental group) vs. usual rehabilitation programs (control group) and assessment at end of treatment and six months after treatment.

The aim of the treatment will be the prevention of falls.

ELIGIBILITY:
Inclusion Criteria:

Patients with stroke, Parkinson's disease and Multiple Sclerosis residing in the centers' catchment areas, requiring rehabilitation, and releasing a written informed consent.

Exclusion Criteria:

1. Cognitive impairment (Minimental State Examination score <21); 2. Major depression; 3. Severe joint/bone disorder interfering with mobility, 4. Aphasia if interfering with understanding the aims of the study and self-administered tests; 5. relapses in the previous three months (MS); 6. Stroke occurred in least four weeks before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Change of Percentage of fallers | Change from Baseline percentage of fallers at 6 months.
  Each patient was given a fall diary and was followed for six months with telephone contacts for six months. The patient (or, if unavailable, the spouse or an informed caregiver) was inquired on targeted rehabilitation programs received during the follow up, the use of walking aid and any incurred falls, with date, circumstances, underlying cause and related injuries. A fall was defined as an unexpected event where the person inadvertently came to rest on the ground or other lower level subjects with >1 falls in the 6 months follow up were categorized as "faller".

SECONDARY OUTCOMES:
Change of Participation level | Change from Baseline partecipation at 6 months.
  The patient (or, if unavailable, the spouse or an informed caregiver) was inquired on partecipation level.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Gnocchi ONLUS, Milan, Italy